CLINICAL TRIAL: NCT00489619
Title: Safe Pregnancy by Infectious Disease Control in the Democratic Republic of Congo - Pilot Study
Brief Title: Safe Pregnancy by Infectious Disease Control
Status: Completed | Type: Observational
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); University of North Carolina (Other); Kinshasa School of Public Health (Other)
Responsible Party: Sponsor
Other Study IDs: GN 02 - Pilot; U01HD043475 (NIH)
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Pregnancy; Malaria
Keywords: Infectious diseases; Democratic Republic of Congo; Malaria; International; Maternal and child health; Women's Health; Global Network; Sexually transmitted infections (STIs)
MeSH Terms: conditions — Malaria; Communicable Diseases; Sexually Transmitted Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Malaria and sexually transmitted infections (STIs) are common in pregnant women in Africa and are important preventable causes of poor birth outcomes and maternal and infant mortality. This study investigated baseline characteristics of the population including: rates of STIs including HIV, prevalence of malaria and tuberculosis (TB) and resistance to common antimalarial drugs.

DETAILED DESCRIPTION:
A cross-sectional observational study was conducted with 2008 pregnant women attending either Binza or Kingasani Maternity clinics in Kinshasa, DRC to determine baseline rates of STIs, TB and malaria. Data was collected for sample size calculation in a larger STI/Malaria and TB randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* older than or equal to 15 years of age
* pregnant
* presenting for antenatal care at one of the two target maternities for the first time during the current pregnancy
* willing to provide informed consent

Exclusion Criteria:

* refusal to participate in the HIV voluntary and counseling program at the maternity center or refusal to share HIV results with the study staff.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2008 (Actual)
Dates: Start 2004-04; Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Ryder, M.D., Principal Investigator — University of North Carolina
Locations (2):
- Democratic Republic of the Congo (2):
  - Binza Maternity, Kinshasa
  - Kingasani Maternity, Kinshasa

REFERENCES:
- See also: Global Network for Women's and Children's Health Research — http://gn.rti.org
- See also: Research Triangle Institute International — http://www.rti.org